CLINICAL TRIAL: NCT03157843
Title: Rate of Venous Thrombosis in Acutely Ill Patients Hospitalized in Internal Medicine Wards
Acronym: AURELIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Violi, Principal Investigator, Clinical Professor, MD, University of Roma La Sapienza
Other Study IDs: AURELIO
Record Dates: First submitted 2016-10-09; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Venous Thromboembolism; Deep Venous Thrombosis
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Medical Patients: Medical patients who received, at admission and during all the length of recovery, antithrombotic drugs (low-molecular-weight heparin at prophylactic dosage ).
  Interventions: Drug: low-molecular-weight heparin
- Control Group: Medical patients not treated with antithrombotic drugs during the recovery. Subjects age, sex and comorbidities matched.

INTERVENTIONS:
Drug: low-molecular-weight heparin
  Groups: Medical Patients

SUMMARY:
After reports from observational studies suggesting an association between acutely ill medical patients and venous thromboembolism (VTE), interventional trials with anticoagulants drugs have demonstrated a significant reduction of VTE during and immediately after hospitalisation. Although several guidelines suggest the clinical relevance of reducing this outcome, there is a low tendency to use anticoagulants in patients hospitalised for acute medical illness. This observational multicentre study wants to evaluate the incidence of venous thrombo-embolism in acutely ill patients hospitalized in internal medicine wards.

DETAILED DESCRIPTION:
Epidemiological studies have provided evidence of a high rate of thromboembolism in patients hospitalised in medical wards. Based on this, several clinical trials with anticoagulants including low-molecular-weight heparin (LMWH) and fondaparinux have been performed in patients hospitalised for acute medical illness to prevent thromboembolism. Interventional trials consistently showed that prophylaxis with anticoagulants reduces the risk of composite endpoints of deep venous thrombosis (DVT), pulmonary embolism (PE) and DVT-related death. These results prompted recommendation to the use anticoagulant prophylaxis in patients hospitalised for acute medical illness, but, despite this, there is a widespread underuse of anticoagulant prophylaxis in the medical wards of hospitals.

This observational multicentre study wants to evaluate the incidence of venous thrombo-embolism in acutely ill patients hospitalized in internal medicine wards.

ELIGIBILITY:
Inclusion Criteria:

* pneumonia
* heart failure
* Chronic Obstructive Pulmonary Disease
* Kidney failure
* syncope
* atrial fibrillation
* Urinary Tract Infection
* Anemia
* arthritis
* Diabetic Ketoacidosis
* unstable angina
* asthma
* cirrhosis

Exclusion Criteria:

* treatment with vitamin k inhibitors
* surgical interventions
* deep venous thrombosis
* pulmonary embolism

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalised for acute medical illness
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Venous thrombo-embolism | Baseline, up to 4 weeks
  Evaluation of deep venous thrombosis by compression ultrasonography (CUS)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violi, MD, Study Chair — Internal and Medical Specialties Department, Policlinico Umberto I, Rome, Italy, 00161; Lorenzo Loffredo, MD, Study Director — Internal and Medical Specialties Department, Policlinico Umberto I, Rome, Italy, 00161
Locations (1):
- Sapienza University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loffredo L, Vidili G, Sciacqua A, Cogliati C, Di Giulio R, Bernardini S, Ciacci P, Pietrangelo A, Orlando F, Paraninfi A, Boddi M, Di Minno G, Falsetti L, Lodigiani C, Santoliquido A, Ettorre E, Pignatelli P, Arezzo MF, Gutu E, Harenberg J, Violi F; AURELIO Study Group. Asymptomatic and symptomatic deep venous thrombosis in hospitalized acutely ill medical patients: risk factors and therapeutic implications. Thromb J. 2022 Nov 30;20(1):72. doi: 10.1186/s12959-022-00433-8. PMID 36451162